CLINICAL TRIAL: NCT04942587
Title: The Effect Of Lullaby Records Sung By The Parent's During Newborn Care On Newborn's And Physical Parameters In Newborn Intensive Care Unit
Brief Title: The Effect Of Lullaby Records Sung By The Parent's During Newborn Care On Newborn's
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Duygu Akyuz, Principal Investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KÜ GOKAEK 2018/90
Record Dates: First submitted 2021-06-15; First posted 2021-06-28 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Comforf, Procedural (During Newborn Care İn Newborn's); Physiological Parameters During Newborn Care İn Newborn's
Keywords: Mother's voice; Father's voice; Lullaby; Comfort; Physiological Parameters

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mother's voices (Experimental): Standard nursing care including, eye, mouth, nose, diaper change, skin care with baby oil and nurturing was applied respectively to the study groups for approximately 20 minutes. The baby was made listen to the lullaby recorded in the voice of mother's starting with, during and after the care for 10 minutes. Heart rate, saturation, respiration rate and comfort behiavour scores of the newborn was measured 1 minutes before, during and 15 minutes after the care.
  Interventions: Behavioral: LISTENING TO THE RECORDINGS SAYING BY PARENTS
- father's voices group (Experimental): Standard nursing care including, eye, mouth, nose, diaper change, skin care with baby oil and nurturing was applied respectively to the study groups for approximately 20 minutes. The baby was made listen to the lullaby recorded in the voice of father's starting with, during and after the care for 10 minutes. Heart rate, saturation, respiration rate and comfort behiavour scores of the newborn was measured 1 minutes before, during and 15 minutes after the care.
  Interventions: Behavioral: LISTENING TO THE RECORDINGS SAYING BY PARENTS
- control group (No Intervention): Standard nursing care including, eye, mouth, nose, diaper change, skin care with baby oil and nurturing was applied respectively to the study groups for approximately 20 minutes.Heart rate, saturation, respiration rate and comfort behiavour scores of the newborn was measured 1 minutes before, during and 15 minutes after the care.

INTERVENTIONS:
Behavioral: LISTENING TO THE RECORDINGS SAYING BY PARENTS — The baby was made listen to the lullaby recorded in the voice of parents starting with, during and after the care for 10 minutes.
  Arms: father's voices group; mother's voices

SUMMARY:
Standard nursing care including, eye, mouth, nose, diaper change, skin care with baby oil and nurturing was applied respectively to the study groups for approximately 20 minutes. The baby was made listen to the lullaby recorded in the voice of parents starting with, during and after the care for 10 minutes. Heart rate, saturation, respiration rate and comfort behiavour scores of the newborn was measured 1 minutes before, during and 15 minutes after the care. The data was evaluated in SPSS 21.0 program with convenient statistical methods.İt is detected that heart rate, respiration rateand comfort behiavour scores of the newborns who listen to lullaby in the mother's voice are low compared to the newborns listening to lullaby in the father's voice and those in the control group .

ELIGIBILITY:
Inclusion Criteria:

* Premature babies at 30-37 weeks of gestation,
* There is no congenital anomaly affecting respiration and spontaneous respiration,
* No intubation,
* Absence of congenital or acquired malfarmation related to hearing,
* Absence of hyperbilirubinemia requiring exchange transfusion,
* Absence of intrauterine infection (rubella, syphilis, toxoplasma),
* Absence of intracranial bleeding,
* No sedative, opioid and anticonvulsant drugs were given before/during the study,
* Parents' consent to participate in the study,

Exclusion Criteria:

* Having a diagnosis of asphyxia,
* Congenital hearing problems in family members,
* Intubating the baby after starting the research,
* Parents have a speech impediment,
* Parents have psychological problems,

Ages: 30 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2019-01-20 (Actual)

PRIMARY OUTCOMES:
The effect of lullaby records sung by the parent's during newborn care on newborns comfort in newborn intensive care unit. | 35 minute
  Newborn comfort behavior scale was used for determinain Comfort behiavour scores in this research. Scale got 0 to 35 points (0 (Good) to 35 (Bad).
The effect of lullaby records sung by the parent's during newborn care on newborns on the heart beat in newborn intensive care unit. | 35 minute
  heart beat- bpm
The effect of lullaby records sung by the parent's during newborn care on newborns on the respiration rate in newborn intensive care unit. | 35 minute
  respiration rate
The effect of lullaby records sung by the parent's during newborn care on newborns on the SpO2 in newborn intensive care unit. | 35 minute
  ects of the use of baby mobile accompanied with Brahms Lullaby on the baby's SpO2 during sternum dressing SpO2

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Akyüz, Principal Investigator — binayduygu@gmail.com; Gülzade Uysal, Principal Investigator — gülzadeuysal@gmail.com
Locations (1):
- University of Kocaeli Hospital, Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes